CLINICAL TRIAL: NCT00034463
Title: A Phase 1 Trial of ALIMTA (Pemetrexed) in Patients With Locally Advanced or Metastatic Cancer
Brief Title: ALIMTA (Pemetrexed) in Patients With Locally Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 1310; H3E-MC-JMAS
Record Dates: First submitted 2002-04-29; First posted 2002-04-30 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Metastases; Cancer
Keywords: metastatic cancer; chemotherapy
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — Pemetrexed; Folic Acid

INTERVENTIONS:
Drug: ALIMTA
Drug: folic acid
Drug: multi-vitamins

SUMMARY:
This is a non-randomized, phase 1, study with the primary objective of determining the toxicities and establishing the maximum tolerated dose of ALIMTA when administered as a 10 minute infusion every 21 days with folic acid or multi-vitamin supplementation therapy in lightly or heavily pre-treated patients with locally advanced or metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of metastatic or locally advanced cancer
* Prior chemotherapy is allowed
* Adequate bone marrow, liver and kidney function

Exclusion Criteria:

* Prior treatment with ALIMTA
* Brain metastasis
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., San Antonio, Texas, United States